CLINICAL TRIAL: NCT05916001
Title: Multicenter RCT on Effects of Preoperative Immunonutrition on Patients Undergoing Elective Colorectal Surgery for Neoplasm: Changes in Adipose Tissue Inflammation and Correlation With Surgical Outcome for Future ERAS Guidelines.
Brief Title: Preoperative Immunonutrition in Patients Undergoing Elective Colorectal Surgery for Neoplasm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giuseppe Nigri, MD, PhD, FACS, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 7064/2023
Record Dates: First submitted 2023-03-15; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Cancer of Colon; Nutrition Related Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A, Impact oral + Colorectal Surgery (Active Comparator): the supplement Oral Impact will be administered 3 times a day for 10 days before the operation.
  Colon surgery will be performed according to standard clinical practice.
  Interventions: Dietary Supplement: Oral Impact Nestle; Procedure: Colorectal surgery
- B, Placebo group + Colorectal Surgery (Placebo Comparator): A Placebo will be administered 3 times a day for 10 days before the operation. Colon surgery will be performed according to standard clinical practice.
  Interventions: Other: Placebo; Procedure: Colorectal surgery

INTERVENTIONS:
Other: Placebo — A Placebo will be administered per os 3 times per day for 10 days before colorectal surgery
  Arms: B, Placebo group + Colorectal Surgery
Dietary Supplement: Oral Impact Nestle — Oral Impact Nestle will be administered per os 3 times per day for 10 days before colorectal surgery
  Arms: A, Impact oral + Colorectal Surgery
Procedure: Colorectal surgery — Colorectal surgery will include right colectomy, left colectomy, transverse colectomy, anterior rectal resection. All procedures will be performed according to the standard clinical practice.

SUMMARY:
Enhanced Recovery After Surgery (ERAS) protocols were developed to standardize perioperative practice in colon surgery to reduce morbidity, improve recovery, and shorten length of stay (LOS). Better protocol adherence translates into fewer readmissions and complications, and better 5-year survival. Preoperative elements, especially nutrition and immunonutrition, are topics that need further development to become the standard of care. It has been widely reported that the prevalence of malnutrition reaches 40% in cancer patients at the time of diagnosis. Impaired nutritional status at the time of surgery and cancer-induced inflammation, along with postoperative inflammatory responses to major surgery, increase the risk of postoperative complications, along with a decrease in perceived quality of life.

Immunonutrition can modulate inflammation and reduce postoperative infections and shorten length of stay by counteracting the immune response induced by cancer. Adipose tissue has been shown to be a relevant source of inflammatory mediators, which may play a role in the promotion of tumor cachexia.

The present study is a multicenter randomized control study (RCT) designed to evaluate the effect of preoperative immunonutrition in patients with colorectal cancer eligible for elective minimally invasive procedures, evaluating in particular surgical site infection and length of hospital stay. A biopsy of subcutaneous adipose tissue and visceral adipose tissue will also be performed, in order to evaluate the differences between inflammatory infiltrate, degree of fibrosis and cross-sectional area of adipocytes compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* primary colorectal neoplasms eligible for elective surgery, undergoing minivasive resections.
* 20 to 85 years old, with no difficulties in oral intake
* BMI ranging from 18 to 40.

Exclusion Criteria:

* emergency surgery,
* converted procedures,
* major intraoperative complications,
* concomitant chronic disease such as chronic renal failure, rheumatic and hematological disease, chronic inflammatory bowel diseases,
* synchronous cancer,
* previous bowel resections or bariatric surgery,
* presence of preoperative stoma.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection (SSI) | 30 days after the surgical procedure
  Number of participants developing surgical site infections (SSI), defined as wound/parietal infection or intra-abdominal abscess without any anastomotic leak.

SECONDARY OUTCOMES:
Anastomotic leakage (AL) | 30 days after the surgical procedure
  Number of participants developing anastomotic leakage (AL), defined as the evidence of leakage at the ileocolic or colo-colic or colo-rectal anastomosis, diagnosed with imaging modalities or with reoperation
Length of stay (LOS) | at patients' discharge
  Mean and Median Length of stay (LOS), defined as the mean and median number of days of hospitalization from the day of the surgical procedure to the day of patients' discharge
Inflammatory infiltration in the subcutaneous adipose tissue (SAT) and visceral adipose tissue (VAT) | at the time of tissue analysis, usually 1 month after surgery
  Number of inflammatory cells in the specimens of subcutaneous adipose tissue (SAT) and visceral adipose tissue (VAT), as stated in a previous study published by the investigators (Molfino A, J Cachexia Sarcopenia Muscle. 2022 Feb;13(1):333-342.).
grade of fibrosis in the subcutaneous adipose tissue (SAT) and visceral adipose tissue (VAT) | at the time of tissue analysis, usually 1 month after surgery
  Number of fibroblasts in the specimens of subcutaneous adipose tissue (SAT) and visceral adipose tissue (VAT), as stated in a previous study published by the investigators (Molfino A, J Cachexia Sarcopenia Muscle. 2022 Feb;13(1):333-342.).
Adipocytes cross sectional area (CSA) in the subcutaneous adipose tissue (SAT) and visceral adipose tissue (VAT) | at the time of tissue analysis, usually 1 month after surgery
  Adipocytes cross sectional area (CSA) in the specimens of subcutaneous adipose tissue (SAT) and visceral adipose tissue (VAT), as stated in a previous study published by the investigators (Molfino A, J Cachexia Sarcopenia Muscle. 2022 Feb;13(1):333-342.).